CLINICAL TRIAL: NCT02663375
Title: Symetis ACURATE TA™ Valve Implantation Using TransApical Access:SAVI2 Registry
Brief Title: ACURATE TA™ Valve Implantation Registry: SAVI 2
Acronym: TA-SAVI2
Status: Completed | Type: Observational
Sponsor: Symetis SA (Industry)
Responsible Party: Sponsor
Organization: Boston Scientific Corporation (Industry)
Other Study IDs: 2013-04
Record Dates: First submitted 2014-12-08; First posted 2016-01-26 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Aortic Stenosis
Keywords: TAVI; Aortic Stenosis; Transcatheter aortic valve replacement; Transcatheter aortic valve implantation; Transapical Access
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ACURATE TA™ Transapical Aortic Biorposthesis: Patients implanted with ACURATE TA™ Transapical Aortic Biorposthesis and Delivery System
  Interventions: Device: ACURATE TA™ Transapical Aortic Bioprosthesis

INTERVENTIONS:
Device: ACURATE TA™ Transapical Aortic Bioprosthesis — ACURATE TA™ Transapical Aortic Bioprosthesis is intended for subjects with severe symptomatic aortic stenosis and are considered high risk for surgical conventional Aortic Valve Replacement.
  Other Names: ACURATE TA™ Transapical Aortic Bioprosthesis and delivery System

SUMMARY:
Post-market registry on ACURATE TA™ Transapical Aortic Bioprosthesis and ACURATE TA™ Delivery System implantation in patients presenting severe symptomatic aortic stenosis to collect continued surveillance data pertaining to safety and performance of the device.

DETAILED DESCRIPTION:
The SAVI2 registry is a single arm, prospective, multicenter, non-randomized and open registry up to 1 year follow-up with the Symetis ACURATE TA™.

The ACURATE TA™ is an aortic bioprosthesis for minimal invasive implantation via transapical access to treat patients with severe symptomatic aortic stenosis where conventional aortic valve replacement (AVR) via open surgery is considered to be associated with high surgical risk.

The primary objectives of the registry is to further evaluate the safety and performance of the implantation and the safety at 30-Day Follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient has severe aortic stenosis
* Native aortic annulus diameter from ≥ 21mm up to ≤ 27mm
* Patient willing to participate in the study and provides signed EC-approved informed consent
* The subject and treating physician agree the subject will return for all required post-procedure follow-up visits

Exclusion Criteria:

* Patients are excluded from the registry if they are not eligible for transcatheter treatment of severe aortic stenosis with the ACURATE TA™ and Delivery System as per the Instructions For Use.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ACURATE TA™ is approved for use to treat patients with severe aortic stenosis, the inclusion criteria are broad in order to allow the device to be used in an all-comers population and following the Instructions For Use.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Rate of all-cause mortality at 30 days follow-up | 30-Day Follow-up
  Rate of all-cause mortality at 30 days follow-up

SECONDARY OUTCOMES:
Rate of clinical endpoints (VARC II) at 30 days and 12 months | 30-Days and 12 Months Follow-up
  Rate of clinical endpoints (VARC II) at 30 days and 12 months:
  * Mortality
  * Stroke
  * Myocardial infarction
  * Bleeding complication
  * Acute kidney injury
  * Vascular complication
  * Conduction disturbances and arrhythmia
  * Other TAVI-related complications
Procedural success post-implant | Procedure to 24h Post-implantation
  Procedural success post-implant defined as ACURATE TA™ implanted in intended location with the following criteria:
  * Insufficiency < +3
  * Mean aortic gradient < 20 mmHg
  * EOA ≥ 1.0 cm2
  * No valve-in-valve or conversion to surgery performed
Device success at 7 Day or Discharge (which ever comes first) and at 12 months follow-up | 7-Days Follow-up and 12-Months Follow-up
  Device success analyzed by ECHO measurement at 7 days or discharge (whichever occurs first) and at 12 months follow-up and defined as the following criteria:
  * ACURATE TA™ implanted in intended location
  * No impingement of the mitral valve
  * Normal coronary blood flow
  * Valve-in-valve insufficiency < +3
  * Mean gradient < 20mmHg
  * EOA ≥ 1.0 cm2
  * No valve-in-valve or conversion to surgery performed
Functional improvement from baseline as per NYHA Functional Classification at 30 days and 12 months | 30-Day and 12-Month Follow-up
  Functional improvement from baseline as per NYHA Functional Classification at 30 days and at 12 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Walther, Professor, Principal Investigator — Kerckhoff Klinik
Locations (27):
- Wiener Krankensanstaltenverbund Krankenhaus Hietzing mit Neurologischem Zentrum Rosenhügel, Vienna, Austria
- Germany (23):
  - Klinikum Augsburg, Augsburg
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Herz- und Gefäßzentrum Bad Bevensen, Bad Bevensen
  - Kerckhoff-Klinik, Bad Nauheim
  - Herz- und Gefäßklinik GmbH, Bad Neustadt an der Saale
  - Herz- und Diabeteszentrum NRW ,Bad Oeynhausen Klinik für Thorax- und Kardiovaskularchirurgie, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg, Bernau
  - Klinikum der Ruhr-Universität Bochum Klinik für Herz-und Thoraxchirurgie, Bochum
  - Herzzentrum Universitätsklinikum Köln, Cologne
  - Sana-Herzzentrum Cottbus GmbH, Cottbus
  - Technische Universität Dresden, Dresden
  - Klinik für Kardiologie und Thorax-Kardiovaskuläre_Westdeutsches Herzzentrum Essen, Essen
  - Justus-Liebig-Universität Gießen, Giessen
  - Klinik für Thorax-, Herz- und Gefäßchirurgie Georg-August-Universität, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf Klinik für Herz-und Gefässchirurgie, Hamburg
  - Klinik für Herzchirurgie Karlsruhe GmbH, Karlsruhe
  - Herzzentrum Leipzig GmbH, Leipzig
  - Deutsches Herzzentrum München des Freistaates Bayern, München
  - Klinikum Nürnberg Süd, Nuremberg
  - Universitätsklinikum Regensburg Klinik und Poliklinik für Herz-, Thorax- und herznahe Gefäßchirurgie, Regensburg
  - SHG-Kliniken Völklingen Klinik für Herz-, Thorax- und Gefäßchirurgie, Völklingen
  - Universitätsklinikum Würzburg Klinik für Thorax-, Herz- und Thorakale Gefäßchirurgie, Würzburg
- U.O.C. cardiochirurgia per adulti- Stabilimento di Massa, Massa, Italy
- Switzerland (2):
  - Inselspital-Stiftung, Universitätsklinik für Herz- und Gefässchirurgie, Bern
  - Universität Zürich, Universitätsklinik für Herz- und Gefässchirurgie, Universitätsspital, Zurich